CLINICAL TRIAL: NCT03197181
Title: Causal Role of Frontopolar Cortex for Motivation in Healthy Older Adults: a Transcranial Direct Current Stimulation Study
Brief Title: Frontopolar Cortex and Motivation in Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FPC-17-AGING-01
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Motivation in Healthy Older Adults
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: In two separate sessions, participants receive either anodal or sham transcranial direct current stimulation while the participants are performing a decision-making task on the computer.
Who Masked: Participant
Masking Description: The participants are blind to whether the participants receive anodal or sham stimulation in a session.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anodal transcranial direct current stimulation (Experimental): anodal transcranial direct current stimulation (current strength: 1 mA, duration: 20 min) over the frontopolar cortex
  Interventions: Device: transcranial direct current stimulation
- sham transcranial direct current stimulation (Sham Comparator): sham transcranial direct current stimulation (current strength: 1 mA, duration: 0.5 min) over the frontopolar cortex
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Participants receive anodal or sham transcranial direct current stimulation while performing effort-based decision tasks.

SUMMARY:
Motivation represents a core aspect of goal-directed behavior as it determines how much effort individuals are willing to invest to reach their goals. While research on effort-based decision-making focuses mainly on effort preferences in younger adults, loss of motivation might be a key component of the apathetic tendencies frequently seen in older adults. However, an open question refers to which brain mechanisms underlie motivational processes in older adults. The investigators have recently shown that the frontopolar cortex plays a crucial in motivating the exertion of rewarded effort in younger adults. The goal of the current study is to determine whether frontopolar cortex plays a crucial role for motivation also in older adults and may thus be a promising target for improving the motivation deficits in healthy aging. Participants perform computer-based experimental tasks measuring the propensity to exert cognitive or physical effort for monetary rewards. During task performance, participants receive anodal or sham transcranial direct current stimulation (tDCS) over their frontopolar cortex. The study tests whether tDCS over frontopolar cortex allows modulating participants' motivation to engage in rewarded effort.

DETAILED DESCRIPTION:
Motivation represents a core aspect of goal-directed behavior as it determines how much effort individuals are willing to invest to reach their goals. While research on effort-based decision-making focuses mainly on effort preferences in younger adults, loss of motivation might be a key component of the apathetic tendencies frequently seen in older adults. However, an open question refers to which brain mechanisms underlie motivational processes in older adults. The investigators have recently shown that the frontopolar cortex plays a crucial in motivating the exertion of rewarded effort in younger adults (Soutschek et al., 2018, Biological Psychiatry). The goal of the current study is to determine whether frontopolar cortex plays a crucial role for motivation also in older adults and may thus be a promising target for improving the motivation deficits in healthy aging. 30 older participants (65-80 years) perform computer-based experimental tasks measuring the propensity to exert cognitive or physical effort for monetary rewards. During task performance, participants receive 1 mA anodal or sham transcranial direct current stimulation (tDCS) over their frontopolar cortex. The study tests whether tDCS over frontopolar cortex allows modulating participants' motivation to engage in rewarded effort.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-80 years
* Informed consent as documented by signature
* Normal or corrected-to-normal vision
* Cognitive and language ability to understand study content and procedure
* Normal cognitive functioning (assessed by MMST)
* BDI-II score < 20

Exclusion Criteria:

* Negative response to TMS/tDCS in past
* History of seizure
* History of stroke or heart attack
* History of head injury
* Psychiatric or neurological disorder
* Metal in body/head
* Implanted medical products like pacemaker, medical pumps, heart catheter
* Headache
* Tinnitus
* Currently taking medication affecting the central nervous system
* Insufficient sleep in preceding night
* Excessive consumption of alcohol within last 24 hours

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
participants' decisions to exert cognitive or physical effort for monetary rewards | All participants perform this decision-making task in both experimental sessions (i.e., both the anodal and the sham stimulation session) for 20 min while receiving anodal or sham stimulation.
  The project seeks to test the causal role of FPC in discounting of cognitive and physical effort in healthy older adults. For that purpose, participants perform a task on a computer which requires the participants to decide whether the participants are willing to exert cognitive or physical effort for a monetary reward. Participants perform this task both under anodal and under sham stimulation. It is tested whether anodal, relative to sham, stimulation increases participants' willingness to engage in rewarded cognitive or physical effort.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe N Tobler, Prof., Principal Investigator — University of Zurich
Locations (1):
- University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No